CLINICAL TRIAL: NCT02810314
Title: Study of Default Mode Network (DMN) on Patients With Multiple Sclerosis (MS)
Brief Title: Default Mode Network in Multiple Sclerosis
Acronym: CONNECT-15
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, María Luisa Martinez Gines, neurologist, Hospital General Universitario Gregorio Marañon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CONNECT-15
Record Dates: First submitted 2016-06-15; First posted 2016-06-22 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical measures (Experimental): MS patients recruited for this study will complete a resting state functional magnetic resonance image (rs-fMRI) session that will provide information on how DMN network works for each group and all MS patients will also complete a comprehensive neuropsychological battery including cognitive and behavioural tests of interest in MS
  Interventions: Behavioral: neuropsychological battery; Other: resting state functional magnetic resonance image (rs-fMRI)
- Control measures (Other): Healthy participants recruited for this study will complete a resting state functional magnetic resonance image (rs-fMRI) session that will provide information on how DMN network works
  Interventions: Other: resting state functional magnetic resonance image (rs-fMRI)

INTERVENTIONS:
Behavioral: neuropsychological battery — neuropsychological battery including cognitive and behavioural tests
  Arms: Clinical measures
Other: resting state functional magnetic resonance image (rs-fMRI) — rs-fMRI

SUMMARY:
The study will evaluate connectivity regardless whether patients present a clinical type that requires medical treatment. In this point, investigators will include patients with progressive evolution as well as initial forms of the disease (CIS) and properly established forms of multiple sclerosis (MS) in remittent-recidivant (RR) forms. The researches will not focus on medical treatment as some of these clinical forms have no indication for disease modifying drugs.

DETAILED DESCRIPTION:
To date, no clear consensus has been reached related to default mode network (DMN) activity and different clinical types of MS. Due to this controversy on the literature regarding increment and decrement of DMN activity along the natural history of MS evolution, this study aim to add experimental information and more data that might help to disentangle this paradox, also correlating this DMN activity with anatomic and cognitive indexes. The investigators will also introduce a novel experimental design, including a prospective measure of the investigators connectivity and cognitive measures.

In this study, investigators aim to evaluate connectivity regardless whether patients present a clinical type that requires medical treatment. In this point, patients with progressive evolution as well as initial forms of the disease (CIS) will be included and properly established forms of MS in RR forms. Researchers will not focus on medical treatment as some of these clinical forms have no indication for disease modifying drugs. Nevertheless, investigators consider that the study of connectivity is worth regardless their pharmacological treatment.

The investigators also aim to offer data on the natural history of MS evolution for distinct MS type patients and healthy controls, as this study is planned to collect data longitudinally.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnostic following McDonald 2010 diagnosis criteria.
* 18 to 60 years old.
* Consent form signature.

Exclusion Criteria:

* Dementia diagnosis, following Spanish Neurological Society criteria.
* Mayor psychiatric illness.
* Physical or intellectual limitations to successfully perform - neuropsychological evaluation.
* Any other circumstance that may interfere with functional magnetic resonance session.
* Abnormal renal function previous to magnetic resonance image (MRI) session.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change of functional connectivity of default mode network (DMN) | at study entry and after 12 months
  measure is taken with fMRI

SECONDARY OUTCOMES:
Correlate grey matter indexes and cognitive functioning indexes | at study entry and after 12 months
  Two measures will be correlated: baseline and after 12 months
Correlate grey matter indexes and emotional/behavioural indexes | at study entry and after 12 months
  Two measures will be correlated: baseline and after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: María Luisa Martínez-Ginés, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No